CLINICAL TRIAL: NCT05231343
Title: A Prospective Randomized Trial Comparing Dual Mini-Fragment Plating to Single Precontoured Plating of Acute Midshaft Clavicle Fractures: A Pilot Study
Brief Title: Comparing Dual Mini-fragment Plating to Single Precontoured Plating of Acute Midshaft Clavicle Fractures Trial
Acronym: COMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Orthopaedic Trauma Society (Other)
Responsible Party: Principal Investigator, Dr. Ujash Sheth, Orthopaedic Surgeon, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPACT
Record Dates: First submitted 2022-01-13; First posted 2022-02-09 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Clavicle Fracture
Keywords: Orthogonal plating; Hardware removal; Reoperation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual mini-fragment plating (Experimental)
  Interventions: Procedure: Dual Mini-fragment Plating
- Single precontoured plating (Active Comparator)
  Interventions: Procedure: Single Precontoured Plating

INTERVENTIONS:
Procedure: Dual Mini-fragment Plating — Patients randomized to dual mini-fragment plating will undergo clavicle fixation using any configuration of 2.0-mm, 2.4-mm and 2.7-mm limited contact dynamic compression (LC-DCP), locking compression (LCP) or reconstruction plates (i.e., 2.4-mm superior and 2.7-mm anteroinferior). One of the two plates used must be a LC-DCP or LCP plate. Surgeons will contour the mini-fragment plate intraoperatively to fit each patient's anatomy.
  Arms: Dual mini-fragment plating
Procedure: Single Precontoured Plating — Patients randomized to a single plate construct will undergo fixation using an anatomically precontoured (superior or anterior-inferior) clavicle plate.
  Arms: Single precontoured plating

SUMMARY:
The rate of surgical fixation of fractures of the collarbone (i.e., midshaft clavicle) has exponentially increased in recent years; however, the rate of repeat procedures for removal of these implants (i.e., plates) due to irritation remains high. Despite technological advances in implant design, nearly one in four patients with a surgically fixed collarbone ultimately undergoes removal of their implant. More recently, there has been a growing body of literature demonstrating the effectiveness of using two smaller caliber plates, which have been found to have similar rates of implant removal. As such, the proposed randomized clinical trial seeks to be the first level I study to directly compare dual mini-fragment plating of acute displaced midshaft clavicle fractures to single precontoured plating. The investigators hypothesize that dual mini-fragment plating will result in lower rates of reoperation with similar rates of union and complication.

DETAILED DESCRIPTION:
Midshaft clavicle fractures have traditionally been treated non-operatively with immobilization in a sling or a figure-of-eight bandage. Early studies reported a non-union rate of 1% and negligible functional consequence with conservative management. However, the inclusion of pediatric fractures and an absence of modern functional assessments in these studies resulted in an underestimation of non-union rates and overly optimistic clinical outcomes. More recent data has demonstrated a non-union rate of 15% with approximately 30% of patients dissatisfied with their outcome following non-operative treatment. As a result, there has been renewed interest in surgical fixation of displaced midshaft clavicle fractures. In fact, the rate of operative fixation has exponentially increased following the publication of a landmark randomized controlled trial by the Canadian Orthopaedic Trauma Society (COTS) which was the first of many level I studies to demonstrate higher union rates, decreased rates of symptomatic malunion, earlier return to function, and improved patient-reported outcomes with plate fixation of displaced midshaft clavicle fractures.

Traditional plating techniques for open reduction and internal fixation of clavicle fractures involved the use of a single 3.5-mm plates placed superiorly or anteriorly. However, these plates are often very prominent under the skin causing irritation, and in many cases result in reoperation for hardware removal. The rate of reoperation for removal of symptomatic hardware has been reported to range from 8% to 66%. For this reason, there have been a number of different fixation strategies describes to minimize the need to return to the operating room for implant-related symptoms. These include intramedullary nailing and the use of anatomic precontoured clavicle plates positioned superiorly or anteroinferiorly. However, even with the use of precontoured plates, the reported hardware removal rate varies from 5% to 47%. This is likely due to the significant variation in clavicle anatomy (i.e., sigmoid curve, coronal bow and length) observed between individuals which precludes anatomic fitting of precontoured plates in all patients. In fact, Malhas and colleagues published a cadaveric study that found further contouring of precontoured plates was necessary in 73% of cases to optimize plate-bone fit.

More recently, a dual plate construct using two mini-fragment plates (i.e., 2.4-mm or 2.7-mm plates) placed orthogonally has been advocated as a means of decreasing the rate of reoperation for symptomatic hardware removal. In 2015, Prasarn et al. reported on a series of 17 patients undergoing clavicle fixation using a 2.7-mm plate positioned superiorly and a 2.4-mm plate positioned anteriorly and had no reoperations while noting a 100% union rate. The idea of dual plating is not new and is commonly used in the setting of clavicle fracture non-union fixation. Its efficacy has also been described in distal clavicle fractures. Dual plating may serve as the ideal low-profile implant option to help diminish the high rates of symptomatic implant removal observed with single plating. The benefits associated with a dual plate construct extend beyond a reduction in implant-related soft-tissue irritation. Intraoperatively, dual plating allows for more points of fixation, buttressing of anterior butterfly fragments, mini-fragment plates to be used as washers for multiple lag screws, and the use of either the superior or anterior plate as a reduction aid or clamp, while the second plate is applied. Based on existing biomechanical data in the literature, the ability of a dual plate construct to withstand multiplanar bending forces better than a single plate construct may also allow for early weight-bearing through the affected extremity. Despite the aforementioned benefits of dual plate fixation, there remains a lack of level I evidence for its use in the surgical management of acute midshaft clavicle fractures.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age
* A completely displaced midshaft fracture of the clavicle (no cortical contact between the main proximal and distal fragments (AO/OTA 15.2A/B/C)
* Fracture amenable to plate fixation with a minimum of three screws in each proximal and distal fragment

Exclusion Criteria:

* Open fracture
* Pathological fracture
* Fracture seen > 28 days after injury
* Associated neurovascular injury
* Associated head injury (Glasgow Coma Scale < 12)
* Concomitant ipsilateral upper extremity fracture
* Significant medical comorbidities (i.e., ASA grade IV and V)
* Inability to comply with follow-up and
* Lack of consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Removal of hardware at two years of follow-up | 24 months postop
  The proportion of people that had their clavicle hardware removed by the two year follow-up.

SECONDARY OUTCOMES:
Radiographic union | 6 weeks, 3 months, 6 months, 12 months and 24 months postop
  Complete cortical bridging between the proximal and distal fragments on both views.
Reoperation causes other than hardware removal | 6 weeks, 3 months, 6 months, 12 months and 24 months postop
  The proportion of people undergoing reoperation for reasons other than hardware removal.
Adverse events/complications | 6 weeks, 3 months, 6 months, 12 months and 24 months postop
  Any event that necessitates another operative procedure or additional medical treatment. Nonunion will be defined as a lack of radiographic healing with clinical evidence of pain and motion at the fracture site at one year. Complex regional pain syndrome will be diagnosed by the presence of dysesthesia and hyperesthesia extending into the hand of the operative limb, with associated vasomotor changes, skin atrophy and diffuse osteopenia.
Operative duration | Immediately after skin closure
  Time between skin incision to skin closure
Pain as measured by the Numeric Pain Rating Scale (NPRS) | 6 weeks, 3 months, 6 months, 12 months and 24 months postop
  The outcome on the Numeric Pain Rating Scale at the time points listed below. The scale ranges from 0 to 10, with a lower score representing less pain and thus a better outcome.
Functional outcome ASES | 6 weeks, 3 months, 6 months, 12 months and 24 months postop
  Functional outcome as measured by the American Shoulder and Elbow Surgeons (ASES) shoulder score. The score values range from 0 to 100, with a lower score representing greater pain and disability.
Functional outcome DASH | 6 weeks, 3 months, 6 months, 12 months and 24 months postop
  Functional outcome as measure by the Disabilities of the Arm, Shoulder and Hand (DASH) score. The score ranges from 0 to 100, with a lower score representing complete, unrestricted functioning of the upper extremities.
Hardware related symptoms | 3 months, 6 months, 12 months and 24 months postop
  As measured by the Clavicle Hardware Irritation Patient Questionnaires (CHIP-Q). This is a qualitative questionnaire.
Numbers of patients screened and eligible for the study within the recruitment period | Enrollment
  We are interested in understanding how many people are eligible for the study.
Numbers of patients who agree to participate | Through study completion, an average 2 years
  We are interested in understanding how many people agree to participate in the study.
Number of patients who have missed data points or time points | Through study completion, an average 2 years
  We are interested in understanding how many people have missed data points or time points in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ujash Sheth, MD MSc FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No